CLINICAL TRIAL: NCT04436328
Title: Conservative Versus Surgical Treatment of Native Vertebral Osteomyelitis: a Randomized Multicentre Trial
Brief Title: Conservative Versus Surgical Treatment of Native Vertebral Osteomyelitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, Head of septic surgery, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Spine infection treatment
Record Dates: First submitted 2020-06-02; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Vertebral Osteomyelitis; Spondylodiscitis; Surgical Procedure, Unspecified
Keywords: Native vertebral osteomyelitis; Treatment; Spinal implant; Antibiotic therapy
MeSH Terms: conditions — Discitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1), controlled, multicentre explorative trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Experimental): Surgical treatment of native vertebral osteomyelitis followed by antimicrobial therapy
  Interventions: Procedure: Surgical treatment
- Antimicrobial treatment (Active Comparator): No surgical intervention, antimicrobial therapy only
  Interventions: Other: Antimicrobial treatment

INTERVENTIONS:
Procedure: Surgical treatment — Surgical treatment of native vertebral osteomyelitis consisting of debridement, spinal decompression and instrumentation using hardware. Additional standard antimicrobial therapy, according to the pathogen and its antimicrobial susceptibility (intravenous route during first 2 weeks, followed by oral route for additional 4 weeks).
  Arms: Surgical treatment
Other: Antimicrobial treatment — No surgical intervention, antimicrobial therapy only, bed rest or temporary external immobilization of affected spinal segment with orthopedic orthesis. Antimicrobial therapy will be administrated according to the pathogen type and antimicrobial susceptibility, with initial intravenous administration for 2 weeks, followed by oral antibiotics for 4 weeks to complete 6 weeks of total therapy.
  Arms: Antimicrobial treatment

SUMMARY:
The optimal treatment of uncomplicated native vertebral osteomyelitis (NVO) is unknown. While some authors recommend surgical treatment (consisting of spinal debridement, decompression and instrumentation using hardware implantation of hardware), others recommend conservative treatment (with antimicrobial therapy alone). In the proposed randomized controlled multicentric trial, we plan to compare the outcome of conservative vs, surgical treatment of NVO regarding (i) infection outcome (i.e. infection-free proportion of subjects), (ii) functional outcome (pain intensity, spine scores, general mobility, quality of life evaluation), and (iii) socioeconomic impact (direct and indirect costs due to NVO).

A total of 350 subjects will be screened, 300 subjects will be randomized 1:1 into 2 arms: experimental (surgical treatment) and control (conservative treatment). Subjects in both groups will receive pathogen-directed antimicrobial therapy for 6 weeks. Excluded will be patients with acute neurologic impairment, extensive bone destruction, epidural/intraspinal abscess and with spinal hardware.

The clinical impact of this study is enormous since it will generate evidence for rational treatment guidelines. We hypothesize that the conservative treatment of uncomplicated NVO is non-inferior to surgical therapy regarding infection outcome. If the conservative treatment of NVO demonstrate non-inferiority, patients may benefit from avoiding unnecessary surgical intervention.

DETAILED DESCRIPTION:
INTRODUCTION AND EVIDENCE. Native vertebral osteomyelitis (NVO) is mainly caused by hematogenous spread from a distant infection focus (e.g. respiratory, urogenital, intestinal tract, oral cavity, skin or intravascular device), typically involving the intervertebral disc space and adjacent vertebral bodies ("spondylodiscitis"). Rarely NVO develops after percutaneous injection or intervention in the spine region without hardware implantation. Recalcitrant back pain unresponsive to conservative measures along with increased systemic inflammatory biomarkers (C-reactive protein) and/or fever or chills is the initial manifestation prompting additional investigations such as collecting blood cultures and spine imaging. Nevertheless, NVO is often diagnosed late or the diagnose is missed, which has a high impact on patient morbidity and mortality, life quality and healthcare costs (prolonged hospital stay, surgical intervention, antimicrobial therapy). Unrecognized primary infection focus causing NVO may lead to further hematogenous spread, potentially affecting other organs, joints and heart valves. The annual incidence of NVO is reported at 5.78 per 100.000 per year and is increasing in the past decades due to aging population, rise of immunocompromised patients and more invasive treatments. The incidence also increased, in part, due to improvements in diagnostic possibilities, including imaging and non-culture-based microbiological techniques. The mortality of NVO ranges between 5 and 20 %, depending on the primary infectious focus, causing pathogen and patient comorbidities.

The treatment goal of NVO is pain relief, prevention or reversion of neurologic deficits, eradication of infection, and establish spinal stability. The indication for conservative versus surgical treatment of uncomplicated NVO (no relevant abscesses, no neurologic impairment, no spine instability) are not uniform and largely depend on institutional/ regional /national preferences, traditions or random choice. A recent systematic review identified only three studies that comparing conservative to surgical treatment. All three studies are retrospective in design. The indication for surgical treatment in the first two studies was neurologic impairment, extensive bone destruction, epidural abscess formation, and failure of non-operative treatment or intractable back pain. These studies reported the complications and reoperation rates, but no formal statistical analysis was performed, in particular the long-term outcome of both treatment modalities is lacking. Other authors (Nastro et al.) treated with orthesis or spinal instrumentation and found no significant differences in both groups after 9 months. No study so far used uniform definition and stratification criteria for infection, neither used a standardized antimicrobial therapy, allowing to evaluate the outcome on the pathogen, pathogenesis, or primary focus of infection. Therefore, evidence-based data is missing to develop rational treatment guidelines for optimal treatment of NVO.

We hypothesize that the conservative treatment of uncomplicated NVO is non-inferior to surgical therapy regarding infection outcome.

AIM. The aim of this multicenter, randomized, controlled study is to compare the long-term outcome including the proportion of infection-free subjects, functional outcome and socioeconomic outcome between conservative and surgical treatment approaches providing novel high-class evidence to resolve this unknown.

MATERIAL AND METHODS. A total of 350 subjects from 8 different centers (Berlin, Munich, Dresden, Leipzig, Jena, Bonn, Magdeburg, Aachen, Cologne, Hamburg) will be screened. With 8 participating study sites, 200 patients are expected to be randomized per year. With a recruitment period of two years (i.e. 400 patients) and a dropout rate of 15%, 140 patients could be analyzed regarding the primary endpoint at 12 months.

Included patients will be randomized 1:1 into 2 arms: surgical arm and conservative arm. Randomization should avoid selection bias for each group. Allocation of treatments will be performed by a computer-generated list. Randomization will be stratified by center. To ensure balanced group sample sizes in the course of patient recruitment, blockwise randomization with varying block sizes will be conducted within the centers. An independent review committee reviews possible failure cases.

1. SURGICAL ARM: Surgical treatment of native vertebral osteomyelitis consisting of debridement, spinal decompression and instrumentation using hardware. Additional standard antimicrobial therapy, according to the pathogen and its antimicrobial susceptibility (intravenous route during first 2 weeks, followed by oral route for additional 4 weeks).
2. CONSERVATIVE ARM: No surgical intervention, antimicrobial therapy only, bed rest or temporary external immobilization of affected spinal segment with orthopedic orthesis. Antimicrobial therapy will be administrated according to the pathogen type and antimicrobial susceptibility, with initial intravenous administration for 2 weeks, followed by oral antibiotics for 4 weeks to complete 6 weeks of total therapy.

Follow-up will be performed 3, 6 and 12 months after surgery (experimental group) or start of antimicrobial therapy (control group).

STATISTICAL ANALYSIS. For analysis of the primary endpoint (proportion of infection-free subjects in both intervention groups one year after treatment initiation), a continuity corrected chi-squared test will be performed at significance of α=0.05. The Log-rank test (two-sided) will be performed and visualized by Kaplan-Meier method. Potential confounders will be considered by using a Cox proportional-hazards regression model. The primary analysis will be conducted following the intention-to-treat (ITT) principle. The number of patients lost to follow up is assumed to be about 15% and will be replaced. Secondary analyses based on the per-protocol and the as-treated participants will be performed. A logistic regression model will be fit to identify prognostic factors for treatment failure by application of resampling techniques for variable selection. We expect a compliance of taking oral antibiotics as prescribed of about 80%. The incompliance is expected to be equally distributed between both groups and should therefore not represent a bias.

ETHICAL CONSIDERATIONS. As both treatment options are considered part of daily practice, a comparative study between both treatment options should be considered as ethically justifiable. However, ethical concerns in both directions are possible. The surgical treatment may be associated with additional surgical-related complications, whereas the conservative treatment group (antimicrobial treatment alone) may be associated with higher treatment failure rate. The Principle Investigator and the Data Monitoring and Safety Board (DMSB) will analyze the intermediate reports and take appropriate actions, if necessary.

STRATEGIES FOR DATA HANDLING. An electronic Case Report Form (eCRF) will be used for data collection. Regular back-up of the database will be performed. The study database is protected by an authentication method. The database will be accessible anytime to the monitor organization and Data Management and Safety Board (DMSB). Data protection is guaranteed by study software: this generates automatically for each patient a pseudonym, consisting of a combination of alphanumeric characters. All study data will be saved in a pseudonymized way. The patient identification list will be stored only locally by each study center.

TRIAL EXPERTISE. The interdisciplinary spine center at Charité has developed into a leading orthopedic and neurosurgical spine centers, certified by the German Spine Society (DWG). The high-volume clinical workload (>10.000 spinal surgeries in the past 5 years) is utilized for extensive training and research, in particular in the field of diagnosis and treatment of spinal infection. Several multicenter IIT´s were initiated by the interdisciplinary septic team.

TRIAL-SUPPORTING FACILITIES. The support will be provided by the coordinating Center for clinical trials, a member of the German network of coordinating centers for clinical trials (KKS). In addition, the trial is supported by the spine section of the German association of Neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years with NVO, diagnosed by microbiology (positive blood culture or vertebral tissue culture) or histopathology.
* Subjects are willing to participate in the study (signed informed consent) and comply with planned follow-up assessments at 3, 6 and 12 months).

Exclusion Criteria:

* Infection due to Mycobacterium spp. or Brucella spp.
* Infection associated with spinal hardware
* Acute neurologic impairment
* Extensive defect of vertebral body (>2 cm)
* Extensive epidural abscess (>1 cm) or intraspinal abscess (any size)
* Spinal instability/deformity requiring immediate stabilisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of infection-free subjects | 12 months after treatment initiation
  Treatment success: Infection-free status defined as (i) absence of clinical signs of native vertebral osteomyelitis (fever, local signs at surgical site), (ii) normal laboratory findings (serum C-reactive protein), (iii) absence of radiological signs of active native vertebral osteomyelitis (progressive bone destruction, implant loosening or migration), and (iv) absence of unplanned surgical interventions or additional antimicrobial treatment.
  Confirmed failure: Persistence or relapse of infection due to the same pathogen.
  Possible failure: Subjects not fulfilling the criteria for treatment success but have no diagnosis of persistence or relapse of native vertebral osteomyelitis

SECONDARY OUTCOMES:
Functional outcome regarding pain intensity | 12 months after treatment initiation
  Pain intensity according to the numerical rating scale (NRS) for the indication of the perceived pain. Values are from 0 (no pain) to 10 (greatest pain imaginable)
Functional outcome regarding mobility according to Nurick scale | 12 months after treatment initiation
  Nurick scale: A six grade system (0-5) based on the difficulty in walking:
  Grade 0: signs or symptoms of root involvement but without evidence of spinal cord disease Grade 1: signs of spinal cord disease but no difficulty in walking. Grade 2: slight difficulty in walking which does not prevent full-time employment Grade 3: difficulty in walking which prevented full time employment or the ability to do all housework, but which was not so severe as to require someone else's help to walk Grade 4: able to walk only with someone else's help or with the aid of a frame. Grade 5 : chairbound or bedridden.
Functional outcome regarding mobility according Oswestry Disability Index | 12 months after treatment initiation
  The Oswestry Disability Index (ODI) will be used in patients with low back pain.
  There are 10 questions to evaluate how the back or leg pain is affecting the patient's ability to manage in everyday life.
  Scoring Method Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score.
  Interpretation 0%-20%: Minimal disability 20%-40% Moderate disability 40%-60%: Severe disability 60%-80%: Crippled 80%-100%: These patients are either bed-bound or exaggerating their symptoms
Functional outcome regarding quality of life using EuroQOL score | 12 months after treatment initiation
  EuroQOL questionnaire is a measure of both clinical and economic value in health care.
  It consists of a descriptive system and a visual analogue scale (EQ VAS). The descriptive system has 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The visual analogue scale has 3 levels of severity (no problems, some problems, extreme problems).
Functional outcome regarding quality of life using SF-36 questionnaire | 12 months after treatment initiation
  The questionnaire is composed of 36 questions organized in eight scales:
  physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and general mental health. Respondents rate each activity on a three-level scale (a lot, a little, not at all). Item responses are then summed with results expressed on a scale ranging from 0 to 100, representing higher values a better function.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berbari EF, Kanj SS, Kowalski TJ, Darouiche RO, Widmer AF, Schmitt SK, Hendershot EF, Holtom PD, Huddleston PM 3rd, Petermann GW, Osmon DR. Executive Summary: 2015 Infectious Diseases Society of America (IDSA) Clinical Practice Guidelines for the Diagnosis and Treatment of Native Vertebral Osteomyelitis in Adults. Clin Infect Dis. 2015 Sep 15;61(6):859-63. doi: 10.1093/cid/civ633. PMID 26316526
- [Result] Bernard L, Dinh A, Ghout I, Simo D, Zeller V, Issartel B, Le Moing V, Belmatoug N, Lesprit P, Bru JP, Therby A, Bouhour D, Denes E, Debard A, Chirouze C, Fevre K, Dupon M, Aegerter P, Mulleman D; Duration of Treatment for Spondylodiscitis (DTS) study group. Antibiotic treatment for 6 weeks versus 12 weeks in patients with pyogenic vertebral osteomyelitis: an open-label, non-inferiority, randomised, controlled trial. Lancet. 2015 Mar 7;385(9971):875-82. doi: 10.1016/S0140-6736(14)61233-2. Epub 2014 Nov 5. PMID 25468170
- [Result] Shiban E, Janssen I, Wostrack M, Krieg SM, Ringel F, Meyer B, Stoffel M. A retrospective study of 113 consecutive cases of surgically treated spondylodiscitis patients. A single-center experience. Acta Neurochir (Wien). 2014 Jun;156(6):1189-96. doi: 10.1007/s00701-014-2058-0. Epub 2014 Mar 27. PMID 24671549
- [Result] Murillo O, Grau I, Lora-Tamayo J, Gomez-Junyent J, Ribera A, Tubau F, Ariza J, Pallares R. The changing epidemiology of bacteraemic osteoarticular infections in the early 21st century. Clin Microbiol Infect. 2015 Mar;21(3):254.e1-8. doi: 10.1016/j.cmi.2014.09.007. Epub 2014 Oct 12. PMID 25618436
- [Result] Rutges JP, Kempen DH, van Dijk M, Oner FC. Outcome of conservative and surgical treatment of pyogenic spondylodiscitis: a systematic literature review. Eur Spine J. 2016 Apr;25(4):983-99. doi: 10.1007/s00586-015-4318-y. Epub 2015 Nov 19. PMID 26585975
- [Result] Valancius K, Hansen ES, Hoy K, Helmig P, Niedermann B, Bunger C. Failure modes in conservative and surgical management of infectious spondylodiscitis. Eur Spine J. 2013 Aug;22(8):1837-44. doi: 10.1007/s00586-012-2614-3. Epub 2012 Dec 18. PMID 23247861
- [Result] Zimmerli W. Clinical practice. Vertebral osteomyelitis. N Engl J Med. 2010 Mar 18;362(11):1022-9. doi: 10.1056/NEJMcp0910753. No abstract available. PMID 20237348